CLINICAL TRIAL: NCT03035084
Title: Is Vitamin D2 Treatment-associated Decrease in 25(OH)D3 Level a Reciprocal Phenomena? A Randomized Controlled Trial
Brief Title: Is Vitamin D2 Treatment-associated Decrease in 25(OH)D3 Level a Reciprocal Phenomena?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: RAC2161235
Record Dates: First submitted 2017-01-15; First posted 2017-01-27 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Vitamin D Deficiency; 25-Hydroxyvitamin D Concentration
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Ergocalciferols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group-2-D3 (Experimental): Subjects with total 25(OH)D more= 20 nmol/l and less= 40 nmol/l will receive vitamin D2 then randomly assigned to vitamin D3
  Interventions: Drug: Vitamin D3; Drug: Vitamin D2
- Group-2-Placebo (Placebo Comparator): Subjects with total 25(OH)D more= 20 nmol/l and less= 40 nmol/l will receive vitamin D2 then randomly assigned to placebo oral capsule.
  Interventions: Drug: Vitamin D2; Drug: Placebo oral capsule
- Group-1-D2 (Experimental): Subjects with 25(OH)D3 more= 40 nmol/l and total 25(OH)D less= 65 nmol/l will be randomly assigned to vitamin D2.
  Interventions: Drug: Vitamin D2
- Group-1-Placebo (Placebo Comparator): Subjects with 25(OH)D3 more= 40 nmol/l and total 25(OH)D less =65 nmol/l will be randomly assigned to placebo oral capsule.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Vitamin D3 — Single oral dose of 50,000 IU of vitamin D3
  Other Names: cholecalciferol
  Arms: Group-2-D3
Drug: Vitamin D2 — Single oral dose of 50,000 IU of vitamin D2
  Other Names: Ergocalciferol
  Arms: Group-1-D2; Group-2-D3; Group-2-Placebo
Drug: Placebo oral capsule — Placebo oral capsule
  Arms: Group-1-Placebo; Group-2-Placebo

SUMMARY:
Several studies have demonstrated that D2 treatment is associated with a decrease in 25(OH)D3 level and therefore have proposed that D3 would be preferable in term of raising total 25(OH)D level. The investigators postulate that the D2 treatment-associated decrease in 25(OH)D3 level may be related to an increase in total 25(OH)D level rather than being specific to D2 treatment, and thus there would be a D3 treatment-associated decrease in 25(OH)D2 level.

The investigators plan to conduct a double-blind placebo-controlled trial to examine the effect of D3 treatment on 25(OH)D2 level and the effect of D2 treatment on 25(OH)D3 leve

ELIGIBILITY:
Inclusion criteria:

* non-pregnant adults (age ≥18 years)
* healthy
* total 25(OH)D level between 20 to 65 nmol/L.
* living in Riyadh area

Exclusion criteria:

* consumption of more than one serving of milk daily
* taking vitamin D supplements
* habitual weekly sun exposure of 10 hours or more
* history of granulomatous, liver, or kidney disease
* taking anticonvulsants, barbiturates, or steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
ANCOVA-adjusted, mean D2-induced change in 25(OH)D3 level group-1 | day 28
ANCOVA-adjusted, mean D3-induced change in 25(OH)D2 level in group-2 | day 28

SECONDARY OUTCOMES:
ANCOVA-adjusted, mean D2-induced change in 25(OH)D3 level group-1 | day 56
ANCOVA-adjusted, mean D3-induced change in 25(OH)D2 level in group-2 | day 56
Pearson correlation between changes in 25(OH)D3 level in the active arm of group-1 and baseline total 25(OH)D level | day 28
Pearson correlation between changes in 25(OH)D2 level in the active arm of group-2 and baseline total 25(OH)D level | day 28
Pearson correlation between changes in 25(OH)D3 level and 25(OH)D2 level in the active arm of each group | day 28

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad M Hammami, MD, PhD, Principal Investigator — King Faisal Specialist Hospital & Research Center (Riydah)
Locations (1):
- King Faisal Specialist Hospital & Research Center, Riyadh, Central, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hammami MM, Abuhdeeb K, Hammami S, Yusuf A. Vitamin-D2 treatment-associated decrease in 25(OH)D3 level is a reciprocal phenomenon: a randomized controlled trial. BMC Endocr Disord. 2019 Jan 18;19(1):8. doi: 10.1186/s12902-019-0337-8. PMID 30658603